CLINICAL TRIAL: NCT06234917
Title: Relieving Peripheral Neuropathic Pain by Increasing the Power-ratio of Low-β Over High-β Activities in the Central Cortical Region With EEG-based Neurofeedback: Study Protocol for a Controlled Pilot Trial
Brief Title: Increasing Sensori-Motor Rhythm Activity by EEG-Neurofeedback to Reduce the Impact of Pain on Daily Functioning
Acronym: SMR-Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut pour la Pratique et l'Innovation en PSYchologie appliquée (Institut Pi-Psy) (Other)
Responsible Party: Principal Investigator, François Vialatte, Director of PiPsy Institute, Institut pour la Pratique et l'Innovation en PSYchologie appliquée (Institut Pi-Psy)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-A00514-35
Record Dates: First submitted 2023-12-12; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Chronic Pain Syndrome; Peripheral Neuropathic Pain
Keywords: EEG; neurofeedback; neuropathic pain; peripheral neuropathy; sensorimotor rhythm; treatment
MeSH Terms: conditions — Neuralgia; Peripheral Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EEG-NFB protocol aimed at increasing the low-β(SMR)/high-β ratio (Experimental): EEG neuromodulation at central (rolandic) cortical level
  Interventions: Other: EEG-based neurofeedback for brain activity modulation
- EEG-NFB protocol aimed at increasing the α(μ)/θ ratio (Active Comparator): EEG neuromodulation at central (rolandic) cortical level
  Interventions: Other: EEG-based neurofeedback for brain activity modulation

INTERVENTIONS:
Other: EEG-based neurofeedback for brain activity modulation — NFB is a type of biofeedback technique for self-modulating brain activities by means of a learning task performed with ongoing sensory (usually visual) feedback to real-time acquisition of either brain imaging or electroencephalographic (EEG) signal, which serves as a biomarker of brain activity

SUMMARY:
Background: Chronic neuropathic pain associated with peripheral neuropathies cannot be attributed solely to lesions of peripheral sensory axons and likely involves alteration in the processing of nociceptive information in the central nervous system in most patients. Few data are available regarding EEG correlates of chronic neuropathic pain. The fact is that effective cortical neuromodulation strategies to treat neuropathic pain target the precentral cortical region, i.e. a cortical area corresponding to the motor cortex. It is not known how these strategies might modulate brain rhythms in the central cortical region, but it can be speculated that sensorimotor rhythms (SMRs) are modified. Another potent way of modulating cortical rhythms is to use EEG-based neurofeedback (NFB). Rare studies previously aimed at relieving neuropathic pain using EEG-NFB training.

Methods/Design: The objective of this single-centre, single-blinded, randomized controlled pilot study is to assess the value of an EEG-NFB procedure to relieve chronic neuropathic pain in patients with painful peripheral neuropathy. A series of 32 patients will be randomly assigned to one of the two following EEG-NFB protocols, aimed at increasing either the low-β(SMR)/high-β ratio (n=16) or the α(μ)/θ ratio (n=16) at central (rolandic) cortical level. Various clinical outcome measures will be collected before and one week after 12 EEG-NFB sessions performed over 4 weeks. Resting-state EEG will also be recorded immediately before and after each NFB session. The primary endpoint will be the change in the impact of pain on patient's daily functioning, as assessed on the Interference Scale of the short form of the Brief Pain Inventory.

Discussion: The value of EEG-NFB procedures to relieve neuropathic pain has been rarely studied. This pilot study will attempt to show the value of endogenous modulation of brain rhythms in the central (rolandic) region in the frequency band corresponding to the frequency of stimulation currently used by therapeutic motor cortex stimulation. In the case of significant clinical benefit produced by the low-β(SMR)/high-β ratio increasing strategy, this work could pave the way for using EEG-NFB training within the armamentarium of neuropathic pain therapy.

DETAILED DESCRIPTION:
1.1 - Description of the research proceedings and study design This is a single-centre, single-blinded, randomized controlled pilot study, in which 32 patients, aged between 18 and 80 years, suffering from painful peripheral neuropathy (DN4 and NRS pain scores ≥4/10), will be randomly assigned to one of the two following EEG-NFB protocols, aimed at increasing either the SMR/high-β ratio (n=16) or the μ/θ ratio (n=16) at central (rolandic) cortical level in a 1:1 allocation ratio, stratified by age and gender. The group allocation of the patients will be performed by one investigator not involved in the EEG-NFB task or clinical assessment. Patients will be recruited in the Clinical Neurophysiology department of the Henri Mondor University Hospital, Créteil, France, where the research will take place.

1.2 - Screening and inclusion visits During a routine medical visit, the study will be explained and proposed to the eligible patients and a letter of information about the protocol will be given to them. After a delay of reflection of at least a week, patients who agree to perform this research will be convened for an inclusion visit. After checking the inclusion/exclusion criteria, the informed consent form will be completed and signed by the participant and duly countersigned by the investigator.

During this visit, clinical assessment based on the fulfillment of different scales and questionnaires will be performed.

At the end of the inclusion visit, the patient will be randomized to either SMR/high-β or μ/θ training and the first EEG-NFB session will be performed.

1.3 - NFB trial The trial phase will consist of 12 EEG-NFB sessions over 4 weeks (on 3 consecutive days for 4 weeks). Each NFB session will last about 20 minutes, starting and ending with a recording of 2 minutes of resting-state EEG with eyes closed to investigate the impact of NFB on raw EEG. The NFB procedure will consist of 10 blocks of 75-second training separated by 15-second resting interval.

1.4 - Final visit and follow-up A visit will take place at the end of the trial, 7 days after the last NFB session. During this visit, subjects will be administered almost the same clinical evaluation that they received at the inclusion visit.

For the responders, defined as a reduction ≥30% of the 7-item Interference BPI score after the EEG-NFB procedure, an attempt to perform a transfer task will be proposed to the patient. From data collected during a semi-structured interview by the investigator on the strategy used by the patient to "succeed the game" during the NFB session, the mental process that the patient will have to use in the transfer task will be defined between the investigator and the patient. The purpose of the transfer task is to allow generalization of EEG-NFB benefit in real life conditions by realizing an NFB-like paradigm in which patients are invited to engage in the same cognitive strategies as for NFB but without presentation of the feedback signal.

The patient will have to perform the transfer task for 20 minutes every morning for three weeks. At the end of the third week, the investigator will make a phone call to the patient to record the 7-item Interference BPI score.

Study plan and measures:

Inclusion visit: Inclusion/exclusion criteria; Signed informed consent; DN4 questionnaire; Randomization; Baseline assessment (BFI-fr, FMI-fr, BIS-fr, CSI, Exp-LoC-Q); Primary clinical outcome measures: BPI; Other clinical outcome measures (NRS, VRS, NPSI, PCS, HAD, TMT, FSS, LSEQ) 10 EEG-NFB sessions (4 weeks): Resting-state EEG recording; EEG-NFB procedure

1 week after the last EEG-NFB session: Primary clinical outcome measures: BPI; Other clinical outcome measures (NRS, VRS, NPSI, PCS, HAD, TMT, FSS, LSEQ); Analgesic response, PGIC, Side effects After 3 weeks of transfer task (for responders to EEG-NFB): Primary clinical outcome measures: BPI

ELIGIBILITY:
Inclusion Criteria:

* Definite peripheral neuropathy on both clinical and neurophysiological grounds, present for at least 6 months.
* Neuropathic pain clearly related to the neuropathy, as defined by a score ≥ 4/10 on the DN4 questionnaire.
* Score ≥ 4/10 on a 0-10 numerical rating scale (NRS) concerning the average intensity of daily ongoing pain.
* Age between 18 and 80 years.
* Affiliation with the social security system.
* Ability to provide signed informed consent.

Exclusion Criteria:

* Neurological disorder other than peripheral neuropathy (neurodegenerative disorders, migraine, epilepsy, stroke, tumor).
* Psychiatric illness.
* Major visual disturbance.

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Interference Scale of the short form of the Brief Pain Inventory (BPI) | From enrollment to 7 days after the last NFB session
  The 7-item Interference Scale of the short form of the Brief Pain Inventory measures how much pain has interfered with seven daily activities, including general activity, walking, work, mood, enjoyment of life, relations with others, and sleep. It uses a 0 to 10 numeric rating scales for each item rating. The minimum score is 0 (no interference of pain on daily living activities, ie better outcome) and the maximum score is 70 (maximal interference of pain on daily living activities, ie worse outcome).

SECONDARY OUTCOMES:
Average intensity of daily ongoing pain on a 0-10 numeric rating scale (NRS) | From enrollment to 7 days after the last NFB session
  The 0-10 numeric rating scale (NRS) measures the average intensity of daily ongoing pain. The minimum score is 0 (no pain, ie better outcome) and the maximum score is 10 (maximal pain, ie worse outcome).
Average intensity of daily ongoing pain on a 0-5 verbal rating scale (VRS) | From enrollment to 7 days after the last NFB session
  The 0-5 verbal rating scale (VRS) measures the average intensity of daily ongoing pain. The minimum score is 0 (no pain, ie better outcome) and the maximum score is 5 (unbearable pain, ie worse outcome).
Symptomatic profile of neuropathic pain on the Neuropathic Pain Symptom Inventory (NPSI) | From enrollment to 7 days after the last NFB session
  The Neuropathic Pain Symptom Inventory (NPSI) measures the neuropathic pain symptoms specifically. The minimum score is 0 (no pain, ie better outcome) and the maximum score is 100 (maximal neuropathic pain symptoms, ie worse outcome).
Tendency to catastrophizing on the Pain Catastrophizing Scale (PCS) | From enrollment to 7 days after the last NFB session
  The Pain Catastrophizing Scale (PCS) measures the tendency of catastrophizing in daily life. The minimum score is 0 (no catastrophism, ie better outcome) and the maximum score is 52 (maximal tendency to catastrophizing, ie worse outcome).
Anxiety and depression on the Hospital Anxiety and Depression scale (HAD) | From enrollment to 7 days after the last NFB session
  The Hospital Anxiety and Depression scale (HAD) measures the severity of anxiety and depression symptoms, with separate subscores for anxiety and depression. For each subscore, the minimum score is 0 (no anxiety or depression, ie better outcome) and the maximum score is 21 (maximal anxiety or depression, ie worse outcome).
Fatigue on the Fatigue Severity Scale (FSS) | From enrollment to 7 days after the last NFB session
  The Fatigue Severity Scale (FSS) measures the severity of fatigue. The minimum score is 0 (no fatigue, ie better outcome) and the maximum score is 63 (maximal fatigue, ie worse outcome).
Quality of sleep on the Leeds Sleep Evaluation Questionnaire (LSEQ). | From enrollment to 7 days after the last NFB session
  The Leeds Sleep Evaluation Questionnaire (LSEQ) measures the quality of sleep. The minimum score is 0 (poor sleep quality, ie worse outcome) and the maximum score is 100 (maximal sleep quality, ie better outcome).
Dominant peak frequency (PF) of the EEG signal in each frequency band (θ, μ, low-β, and high-β) | At each NFB session through study completion, i.e. 4 weeks
  The dominant peak frequency (PF) of the EEG signal is measured in Hz for each frequency band (θ, μ, low-β, and high-β). There is no better or worse outcome. This is a descriptive data.
Absolute power (AP) of the EEG signal in each frequency band (θ, μ, low-β, and high-β) | At each NFB session through study completion, i.e. 4 weeks
  The absolute power (AP) of the EEG signal is measured in µV² for each frequency band (θ, μ, low-β, and high-β). There is no better or worse outcome. This is a descriptive data.
Relative power (RP) of the EEG signal in each frequency band (θ, μ, low-β, and high-β) | At each NFB session through study completion, i.e. 4 weeks
  The relative power (RP) of the EEG signal is measured in % for each frequency band (θ, μ, low-β, and high-β). There is no better or worse outcome. This is a descriptive data.

CONTACTS AND LOCATIONS:
Locations (1):
- Henri Mondor University Hospital, Créteil, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No